CLINICAL TRIAL: NCT05726240
Title: Multicentre Randomized Trial of Ghrelin in Anterior Circulation Ischemic Stroke Treated With Endovascular Thrombectomy. A Randomized Phase 2 Trial
Brief Title: RCT of Ghrelin in Stroke Patients
Acronym: MR GENTLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR GENTLE
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Stroke, Ischemic
Keywords: Endovascular thrombectomy; Ghrelin
MeSH Terms: conditions — Ischemic Stroke | interventions — Ghrelin

STUDY DESIGN:
Intervention Model Description: This will be a phase 2 multicenter clinical trial with random treatment allocation, open label treatment and blinded endpoint assessment (PROBE design). The intervention contrast will be intravenous acylated ghrelin in addition to standard care (intervention group) vs. standard care alone (control group).
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ghrelin treatment (Experimental): Treatment in the intervention group will consist of intravenous acylated ghrelin, 600micrg dissolved in 50cc normal saline, by bolus (short term) infusion in 30 minutes, twice daily, for five days. This treatment will be additional to standard treatment, including intravenous thrombolysis, if indicated.
  Interventions: Drug: Ghrelin
- Standard care (No Intervention): Treatment in the standard group consists of local practices for the treatment of stroke, including intravenous thrombolysis, if indicated.

INTERVENTIONS:
Drug: Ghrelin — Treatment in the intervention group will consist of intravenous acylated ghrelin, 600micrg dissolved in 50cc normal saline, by bolus (short term) infusion in 30 minutes, twice daily, for five days. This treatment will be additional to standard treatment, including intravenous thrombolysis, if indicated.
  Arms: Ghrelin treatment

SUMMARY:
About half of the patients with acute ischemic stroke treated with endovascular thrombectomy (EVT) remain dependent on the help of others or die in the first 90 days. We hypothesize that treatment with ghrelin, started in the first six hours after stroke onset, improves early recovery and long-term functional outcome in these patients. Ghrelin is a naturally occurring hormone and mildly excitatory neurotransmitter also known as the 'hunger hormone.' Treatment with acylated ghrelin consistently improved functional and histological recovery in in vitro and in vivo models of ischemic stroke.

DETAILED DESCRIPTION:
We will include 80 patients with acute ischemic stroke caused by large vessel occlusion of the anterior circulation, eligible for EVT. The study population will be drawn from adult patients with acute ischemic stroke treated with EVT at UMC Utrecht, Rijnstate, MST or Isala.

Treatment in the intervention group will consist of intravenous acylated ghrelin, 600micrg dissolved in 50cc normal saline, by bolus (short term) infusion in 30 minutes, twice daily, for five days. This treatment will be additional to standard treatment, including intravenous thrombolysis, if indicated.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of acute ischemic stroke, caused by intracranial large vessel occlusion of the anterior circulation (distal intracranial carotid artery or middle (M1/proximal M2) cerebral artery) confirmed by neuro-imaging (CTA or MRA),
* treatment with EVT, defined as groin puncture in the angio suite,
* CT or MRI ruling out intracranial hemorrhage,
* a pre-EVT score of at least 10 on the NIHSS,
* age of 18 years or older,
* written informed consent (deferred).

Exclusion Criteria:

* pre-stroke disability defined as mRS ≥ 2,
* life expectancy shorter than one year,
* child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale score | 7 days after stroke onset
  The primary outcome measure is the score on the National Institutes of Health Stroke Scale at seven days (±1) after stroke onset or at discharge, if earlier. The NIHSS is a continuous scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.

SECONDARY OUTCOMES:
Modified Rankin Scale score | 90 days after stroke onset
  The score on the Modified Rankin Scale at 90 days after stroke onset. The mRS is an ordinal hierarchical scale that describes disabilities encountered post stroke, incorporating six categories from 0 (complete recovery) up to and including 5 (severe disability). 'Death' is assigned a score of 6 .
Mortality | 90 days after stroke onset
  Mortality at 90 days
National Institutes of Health Stroke Scale score | 24 hours after stroke onset
  Scores on National Institutes of Health Stroke Scale at 24 hours after stroke onset. The NIHSS is a continuous scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit. The NIHSS is a continuous scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
National Institutes of Health Stroke Scale score | 72 hours after stroke onset
  Scores on National Institutes of Health Stroke Scale at 72 hours after stroke onset. The NIHSS is a continuous scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit. The NIHSS is a continuous scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Telephonic Montreal Cognitive Assessment | 90 days after stroke onset
  Score on the telephone version of the Montreal Cognitive Assessment at 90 days. The MoCA 5-minute protocol consists of 4 subtests examining 5 cognitive domains, including attention, verbal learning and memory, executive functions/language, and orientation. Total scores of the MoCA 5-minute protocol range between 0 and 30 with lower scores indicating a better cognition.
Infarct size | 72 hours after stroke onset
  Infarct size at 72 hours (based on Magnetic resonance imaging measurements)
Blood glucose levels | Days 1-7 after stroke onset
  Blood glucose levels at days 1-7 (or until discharge)
Blood pressure | Days 1-7 after stroke onset
  Blood pressure at days 1-7 (or until discharge)
Body temperature | Days 1-7 after stroke onset
  Body temperature at days 1-7 (or until discharge)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Utrecht, Utrecht
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Omes QPM, van der Veen D, Kersten CJBA, Arntz RM, Filius PMG, van den Wijngaard IR, van der Worp HB, Hofmeijer J. MR GENTLE-multicentre randomised controlled trial of ghrelin in anterior circulation ischaemic stroke treated with endovascular thrombectomy: a phase 2 trial. Trials. 2026 Jan 16. doi: 10.1186/s13063-026-09426-8. Online ahead of print. PMID 41546024